CLINICAL TRIAL: NCT07134972
Title: The Effect of Ozone Treatment on Coronary Flow Reserve in Patients With Heart Failure Having Reduced Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ekrem Bilal Karaayvaz (Other)
Responsible Party: Sponsor-Investigator, Ekrem Bilal Karaayvaz, Assistant Professor, Istanbul University
Organization: Istanbul University (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulU-EBKaraayvaz-1
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure and Reduced Ejection Fraction
Keywords: ozone treatment; heart failure with reduced ejection fraction; coronary flow reserve
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Intervention Model Description: In our study only the heart failure group have taken ozone treatment. But control groups diagnostic findings were used to compare effect of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group was given no treatment or medication. They had normal echocardiography. They had no heart failure or chronic diseases.
- Study Group (Experimental): Heart failure patients with reduced ejection fraction was administered ozone treatment and diagnosed before and after the treatment to understand ozone treatment's effect.
  Interventions: Drug: Ozone treatment

INTERVENTIONS:
Drug: Ozone treatment — Ozone treatment was administered to study group only. 90 ml of blood was collected into a vacuum sterile glass bottle (Ozonosan). To prevent clotting, 10 ml of 3.8% Na Citrate solution was added to the glass vial. The blood to citrate volume ratio is 9:1. After blood collection, the O3 concentration is ozonized to 20-50 mcg/ml. After at least 5 minutes of mixing, ozonized blood was infused over 20 minutes. Ozone/oxygen mixture was administered intravenously. Ozone therapy was administered twice a week for a total of 16 sessions.
  Other Names: Ozone therapy
  Arms: Study Group

SUMMARY:
The goal of this clinical trial is to determine the effect of ozone treatment in heart failurte with reduced ejection fraction. The main questions it aims to answer are:

Does ozone treatment have beneficial effects in heart failure patients? What medical problems do heart failure patients have when taking ozone treatment? Researchers will compare ozone treatment in patients with heart failure to ozone treatment in patients with no heart failure (control group) as well as before and after the ozone treatment in patients with heart failure to see if ozone works to treat heart failure.

Participants will:

Give blood samples Take 6-minute walk test Be perfomed Echocardiography with CFR (Coronary Flow Reserve) Take drug ABC or a placebo every day for 4 months Visit the clinic twice a week for ozone treatment for 2 months Give blood samples (after the ozone treatment) Take 6-minute walk test (after the ozone treatment) Be perfomed Echocardiography with CFR (Coronary Flow Reserve) (after the ozone treatment)

DETAILED DESCRIPTION:
Patients who were previously scheduled for ozone therapy at the ozone therapy clinic of Medicana International Hospital Istanbul for another indication that did not affect the endothelial function of coronary arteries were included in the study. Patients with diseases or conditions that may affect endothelial function such as diabetes mellitus, chronic renal failure, thyroid or liver dysfunction, inflammatory diseases or smoking were excluded. Thirty-eight patients with non-ischemic cardiomyopathy who underwent coronary angiography in the Cardiology Department of Medicana International Hospital Istanbul and had less than 50% stenosis and less than 40% ejection fraction (EF) on transthoracic echocardiography were included in the study. All participants were taking beta-blockers, ACEi and mineralocorticoid receptor antagonists for the treatment of heart failure. A control group of 22 people with similar age, sex and demographic properties and no chronic disease has included to the study.

After the patients were enrolled in the study, blood samples were taken and 6-minute walk test, CFR measurement and transthoracic echocardiography were performed. They were then sent for ozone therapy. Two months later, after ozone therapy, blood samples were taken and 6-minute walk test, CFR measurement and transthoracic echocardiography were performed again.

ELIGIBILITY:
Inclusion Criteria:

* Previosuly known coronary angiography with less than % 50 stenosis
* Echocardiography with ejection fraction of less than % 40
* Patients with previosly planned for ozone treatment for non-chronic disease or conditions

Exclusion Criteria:

* Known chronic diseases or conditions that effect endothelial functions.
* Previosly had acute coronary syndrome or stent implantation or any coronary intervention.
* Smokers

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Number of patients who had acute heart failure. | From start of the treatment to 2 months after the treatment
  The ozone treatment is used for heart failure in this study. If any patient had acute heart failure episode, whether it is drug related or not, that patient can no longer participate in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ekrem Bilal Karaayvaz, Principal Investigator — Istanbul University Istanbul Faculty of Medicine, Department of Cardiology
Locations (1):
- Medicana International Hospital Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request after the manuscript published
Access Criteria: Data of this study will be upload to clinicaltrials.gov after publication of the study
URL: https://clinicaltrials.gov

REFERENCES:
- [Background] Karaayvaz EB, Guz G. Coronary Flow Reserve Changes after Angiotensin Receptor-Neprilysin Inhibitor Treatment in Heart Failure with Reduced Ejection Fraction. Acta Cardiol Sin. 2023 Nov;39(6):871-878. doi: 10.6515/ACS.202311_39(6).20230619C. PMID 38022415
- [Background] Sawyer DB. Oxidative stress in heart failure: what are we missing? Am J Med Sci. 2011 Aug;342(2):120-4. doi: 10.1097/MAJ.0b013e3182249fcd. PMID 21747279
- [Background] Zuchi C, Tritto I, Carluccio E, Mattei C, Cattadori G, Ambrosio G. Role of endothelial dysfunction in heart failure. Heart Fail Rev. 2020 Jan;25(1):21-30. doi: 10.1007/s10741-019-09881-3. PMID 31686283
- [Background] Katz SD. Mechanisms and implications of endothelial dysfunction in congestive heart failure. Curr Opin Cardiol. 1997 May;12(3):259-64. doi: 10.1097/00001573-199705000-00007. PMID 9243083
- [Background] Heusch G. Coronary blood flow in heart failure: cause, consequence and bystander. Basic Res Cardiol. 2022 Jan 13;117(1):1. doi: 10.1007/s00395-022-00909-8. PMID 35024969